CLINICAL TRIAL: NCT02169180
Title: A Phase 2 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Subjects With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Participants With Relapsed or Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR104615; PCI-32765MCL2002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma, Mantle-cell
Keywords: Ibrutinib; IMBRUVICA; PCI-32765; JNJ-54179060; Lymphoma, Mantle-cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib (Experimental): Participants will receive ibrutinib capsules 560 milligram (mg) orally, once daily on a 28-day cycle up to 7 cycles or until disease progression (or relapse if the participant achieved a complete response [CR]), unacceptable toxicity, or end of treatment, whichever occurs first.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive ibrutinib capsules 560 milligram (mg) orally, once daily on a 28-day cycle up to 7 cycles or until disease progression (or relapse if the participant achieved a complete response [CR]), unacceptable toxicity, or end of treatment, whichever occurs first.
  Other Names: IMBRUVICA; PCI-32765; JNJ-54179060

SUMMARY:
The purpose of this study is to evaluate overall response rate (ORR) (complete response [CR] rate plus partial response [PR] rate) of ibrutinib (IMBRUVICA™; PCI-32765; JNJ-54179060), as assessed by an Independent Review Committee (IRC), in participants with relapsed or refractory mantle cell lymphoma (MCL-a cancer of the lymph nodes or tissues).

DETAILED DESCRIPTION:
This is a Phase 2, single-arm, open-label (all knew the intervention of study), and multicenter (when more than 1 hospital or medical school team work on a medical research study) study to explore the efficacy, safety and pharmacokinetics (the study of the way a drug enters and leaves the blood and tissues over time) of ibrutinib in Japanese participants with relapsed (the return of a medical problem) or refractory (not responding to treatment) MCL. The study will consist of a Screening Phase of 30 days prior to first dose of study drug followed by treatment Phase and a post-treatment follow-up Phase. Participants will receive ibrutinib 560 milligram (mg) orally, once daily on a 28-day cycle until disease progression (or relapse if the participant achieved a CR), unacceptable toxicity, or study end, whichever occurs first. Treatment Phase will have disease assessments every 8 weeks up to 24 weeks after start of study drug, then every 12 weeks thereafter to assess efficacy up to 2 years after last participant enrolled. Efficacy will primarily be evaluated by ORR. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mantle cell lymphoma ( MCL) must include morphology and expression of either cyclin D1 in association with one B-cell marker (for example, cluster of differentiation [CD] CD19, CD20, or paired box [PAX5]) or evidence of t(11;14) as assessed by cytogenetics, fluorescent in situ hybridization (FISH), or polymerase chain reaction (PCR)
* Received at least 1 prior lines of therapy for MCL (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a greater than 6-month treatment-free interval)
* At least 1 measurable site of disease according to the Revised Response Criteria for Malignant Lymphoma (that is, the site of disease must be greater than 1.5 centimeter [cm] in the long axis regardless of short axis measurement or greater than 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions)
* Have documented failure to achieve at least partial response (PR) with, or documented disease progression after, the most recent anti-MCL treatment regimen
* Eastern Cooperative Oncology Group performance status score of 0 or 1

Exclusion Criteria:

* Prior chemotherapy within 3 weeks, nitrosoureas within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy within 3 weeks, or major surgery within 4 weeks of the first dose of study drug
* Prior treatment with ibrutinib or other Bruton's Tyrosine Kinase (BTK) inhibitors
* More than 5 prior lines of therapy for MCL (separate lines of therapy are defined as single or combination therapies that are either separated by disease progression or by a greater than 6-month treatment-free interval)
* Known central nervous system (CNS) lymphoma
* Woman who is pregnant, breast-feeding, or planning to become pregnant within 1 month after the last dose of study drug or is a man who plans to father a child while enrolled in this study or within 3 months after the last dose of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-08; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Overall Response | Up to 2 years after last participant enrolled
  Overall response is defined as achievement of complete response (CR) or partial response (PR), as assessed by the Independent Review Committee (IRC), based on the Revised Response Criteria for Malignant Lymphoma. CR is: a) disappearance of all detectable disease symptoms and signs; b) lymph nodes and nodal masses must have regressed on computed tomography (CT) to normal size; c) negative positron emission tomography (PET) scan; d) normal sized spleen or liver if enlarged before therapy; d) bone marrow infiltrate must be cleared if would have been involved before treatment; e) no new sites of disease. PR is: a) greater than 50 percent decrease in the sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, splenic and hepatic nodules; b) no increase in the size of other nodes, liver, or spleen, c) no measurable disease in other organs; d) no new sites of disease; e) 1 PET-positive site of disease (required for the CT+PET assessment of PR).

SECONDARY OUTCOMES:
Duration of Response | Up to 2 years after last participant enrolled
  Duration of response is defined as the time from the date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Time to Response | Up to 2 years after last participant enrolled
  Time to response is the time from the date of first dose of study drug until the first date of initial documentation of a response (CR or PR).
Overall Survival (OS) | Up to 2 years after last participant enrolled
  The OS is defined as the time from the date of first dose of study drug to date of death from any cause. If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant will be last known to be alive.
Progression-free Survival (PFS) | Up to 2 years after last participant enrolled
  The PFS is defined as the duration from the date of first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death, whichever comes first.
Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Day 1 up to 30 days after last dose administration
  An AE is any untoward medical occurrence in a participant who will receive study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly.
Area Under the Plasma Concentration-Time Curve From Zero to Last Measurable Concentration (AUC [0-t]) | Predose (0), 1, 2, and 4 hours postdose on Day 1 of Cycle 1 and 2
  The AUC (0-last) is the area under the plasma concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Apparent Clearance (CL/F) | Predose (0), 1, 2, and 4 hours postdose on Day 1 of Cycle 1 and 2
  The CL/F is defined as the apparent total clearance of the drug from plasma after oral administration.
Minimum Observed Plasma Concentration (Cmin) | Predose (0) and 1, 2, and 4 hours postdose on Day 1 of Cycle 1 and Cycle 2
  Minimum Observed Plasma Concentration (Cmin) will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (8):
- Japan (8):
  - Fukuoka
  - Isehara
  - Kobe
  - Kyoto
  - Nagoya
  - Osaka
  - Sendai
  - Tokyo

REFERENCES:
- [Derived] Maruyama D, Nagai H, Fukuhara N, Kitano T, Ishikawa T, Shibayama H, Choi I, Hatake K, Uchida T, Nishikori M, Kinoshita T, Matsuno Y, Nishikawa T, Takahara S, Tobinai K. Efficacy and safety of ibrutinib in Japanese patients with relapsed or refractory mantle cell lymphoma. Cancer Sci. 2016 Dec;107(12):1785-1790. doi: 10.1111/cas.13076. Epub 2016 Nov 25. PMID 27616553